CLINICAL TRIAL: NCT05753930
Title: A Single-arm, Multi-centre Trial to Evaluate Efficacy and Safety of Imlifidase in Highly Sensitised Children (1-17 Years) Receiving a Kidney Transplant With Positive Crossmatch Against a Living or Deceased Donor Converted to Negative After Imlifidase Treatment
Brief Title: Imlifidase Prior to Kidney Transplant in Highly Sensitised Children
Acronym: DINKY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-HMedIdes-21; 2022-500230-28-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplantation in Highly Sensitized Patients
Keywords: Desensitization; Highly sensitized; Positive crossmatch; Unlikely to be transplanted; Kidney transplantation; Deceased donor; Living donor; End-Stage Renal Disease; Paediatric patients; Children; Incompatible transplant
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomised trial in highly sensitized paediatric kidney transplant patients with positive XM against an available DD or LD.
  The rationale for a non-randomised trial in DD kidney transplantation is that there are no other effective or approved desensitisation protocols that would provide a suitable or ethical control.
  The rationale for a non-randomised trial in LD kidney transplantation is that potential control treatments have already been tried unsuccessfully in the patients or such treatments are judged as highly unlikely to succeed based on the breadth and depth of the patients' sensitisation. Treatment with little anticipation of success would expose the patients to unnecessary immunosuppression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imlifidase (Experimental): Imlifidase is administered intravenously as one infusion of 0.25 mg/kg over 15 minutes within 24 hours prior to transplantation.
  Interventions: Drug: Imlifidase

INTERVENTIONS:
Drug: Imlifidase — Imlifidase is an immunoglobulin G (IgG)-degrading enzyme of Streptococcus pyogenes that is highly selective towards IgG. The cleavage of IgG generates one F(ab')2- and one homodimeric Fc-fragment and efficiently neutralizes Fc-mediated activities of IgG.
  Other Names: IdeS, HMED-IdeS

SUMMARY:
The goal of this clinical trial is to learn about the efficacy and safety of imlifidase in highly sensitized paediatric patients, 1-17 years old, with end stage renal disease (ESRD).

The main questions it aims to answer are:

* Does imlifidase treatment result in crossmatch conversion that enables transplantation?
* How is the function of the transplanted kidney?

The participants will be hospitalised in accordance with the normal routines for transplanted patients. The patients will receive medication to prevent rejection of the donor kidney, and because such treatment make the body more vulnerable medications to prevent infections.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo pre-screening to determine eligibility for study entry.

The trial will include highly sensitised ESRD paediatric patients (1-17 years). The patients have previously undergone desensitization unsuccessfully or have an anti-HLA antibody status deemed too difficult to make a successful desensitization using other experimental methods.

A screening visit will take place when an organ offer has been placed for a final check of the patients' eligibility for study participation.

All patients included in the trial will be desensitized with imlifidase to convert the positive XM to negative and then transplanted with either a kidney from a deceased donor (DD) or a living donor (LD).

Patients will be hospitalised in accordance with the normal routines for transplanted patients at each clinic.

Following transplantation, the patients will receive induction therapies, rejection prophylaxis, and maintenance immunosuppressive therapies.

The patients will be closely monitored for any signs of antibody-mediated rejections (AMRs).

The duration of the interventional trial period after an organ has been offered will be 6 months for each patient. The trial includes a follow-up part to collect long-term efficacy and safety data up to 5 years after the transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent obtained from patient/parent/legal guardian/independent witness (depending on patient's age) before any trial-related procedures
2. Highly sensitised patient with panel reactive antibodies (PRA) ≥80%
3. Male or female patient between the age of 1 to 17 years (up to the day before the 18th birthday) at the time of screening
4. Patient with end-stage renal disease (ESRD) and waiting for a renal transplant from a living or deceased donor
5. Patient must be transplantable (including size mismatch) at the time of obtaining informed consent for trial participation
6. Patients who have previously undergone desensitisation unsuccessfully with plasmapheresis/IVIg/anti-CD20 or have an anti-HLA antibody status deemed too difficult to make a successful desensitisation (judgement based on physicians' previous experience with similar patients)
7. Positive crossmatch (XM) test determined by flow cytometry crossmatch (FCXM) and/or complement-dependent cytotoxicity crossmatch (CDCXM) tests against the donor. For the DD patients, if physical XM tests are not practically possible due to lack of time, patients may be included on a virtual crossmatch (vXM) predictive of a positive XM test.
8. Willingness and ability to comply with the protocol as judged by the investigator

Exclusion Criteria:

1. Previous treatment with imlifidase
2. IVIg treatment within 28 days prior to imlifidase treatment
3. Desensitisation treatment(s) within 1 month prior to the current transplantation
4. Hypersensitivity to the active substance (imlifidase) or to any of the excipients and to other immunosuppressive drugs specified in the protocol
5. Ongoing serious infections
6. Present, or history of, thrombotic thrombocytopenic purpura (TTP), or known familial history of TTP
7. At the time of transplantation: severe other condition requiring treatment and close monitoring e.g. cardiac failure ≥ grade 4 (New York Heart Association), unstable coronary disease, active peripheral vascular disease, proven hypercoagulable conditions/events or oxygen dependent respiratory disease
8. Malignancy within 3 years prior to transplantation
9. ABO blood group incompatible transplantations (A2 and A2B kidneys will not be accepted for B recipients)
10. Any other reason that, in the view of the investigator, precludes transplantation
11. Breast feeding or pregnancy, if applicable
12. Woman of fertile age and sexually active without adequate contraceptive measures to avoid pregnancy during the interventional trial period (i.e. up to 6 months after transplantation)
13. Suspicion of Covid-19 infection or positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test
14. Positive serology for human immunodeficiency virus (HIV)
15. Clinical signs of hepatitis B virus (HBV), hepatitis C virus (HCV), cytomegalovirus (CMV), or Epstein Barr virus (EBV) infection
16. Donor with positive serology for HIV, HBV, HCV, CMV or EBV to a patient with negative serology (mismatch serology)
17. Clinically relevant active infection(s) as judged by the investigator
18. Tuberculosis or history of tuberculosis
19. Use of other investigational agents within 5 terminal elimination half-lives prior to the transplantation
20. Contemporaneous participation in medical device studies
21. Known mental incapacity or language barriers precluding patients'/parents'/legal guardians' adequate understanding of the informed consent information and the trial activities
22. Inability by the judgement of the investigator to participate in the trial for any other reason

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with conversion of a positive crossmatch test to negative within 24 hours after start of imlifidase treatment | From start of imlifidase administration to 24 hours
  Immunoglobulins (IgG) including donor specific antibodies (DSAs) are rapidly and efficiently cleaved by imlifidase. A conversion of a positive to a negative XM will enable transplantation.

SECONDARY OUTCOMES:
Renal function up to 5 years after transplantation as assessed by estimated glomerular filtration rate (eGFR) | From pre-dose imlifidase up to 5 years
  eGFR is a measure of kidney function. Reduced kidney function is characterised by a decreased eGFR value.
Renal function up to 5 years after transplantation as assessed by serum/plasma creatinine levels | From pre-dose imlifidase up to 5 years
  Creatinine is a measure of kidney function. Reduced kidney function is characterised by an increased value.
Renal function up to 5 years after transplantation as assessed by serum/plasma cystatin C levels | From pre-dose imlifidase up to 5 years
  Cystatin C is a measure of kidney function. Reduced kidney function is characterised by an increased value.
Renal function up to 5 years after transplantation as assessed by proteinuria | From pre-dose imlifidase up to 5 years
  Proteinuria (protein/creatinine ratio in urine) is a measure of kidney function. Reduced kidney function is characterised by an increased value.
DSA levels up to 5 years after transplantation | From pre-dose imlifidase up to 5 years
  Donor specific antibodies (DSAs) are antibodies in the recipient directed against the transplanted organ.
Graft survival (death censored) up to 5 year after transplantation | From 6 months up to 5 years
Graft failure-free survival up to 5 years after transplantation | From 6 months up to 5 years
Patient survival up to 5 years after transplantation | From 6 months up to 5 years
Frequency of delayed graft function (DGF) | From transplantation up 7 days after transplantation
  DGF is defined as 'Need for dialysis within 7 days of transplantation' in "Delayed graft function in kidney transplantation: developing drugs for prevention, guidance for industry", FDA 2019.
  Frequency of patients having DGF in accordance with this definition will be presented.
Length of DGF | From transplantation up 7 days after transplantation
  DGF is defined as 'Need for dialysis within 7 days of transplantation' in "Delayed graft function in kidney transplantation: developing drugs for prevention, guidance for industry", FDA 2019.
  The duration of DGFs in accordance with this definition will be presented.
Proportion of patients with dialysis dependency up to 5 years after transplantation | From 6 months up to 5 years
Imlifidase Pharmacokinetics (AUC) | From pre-dose imlifidase up to Day 15
  AUC = Area under the imlifidase plasma concentration versus time curve.
Imlifidase Pharmacokinetics (Cmax) | From pre-dose imlifidase up to Day 15
  Cmax = Maximum observed plasma concentration of imlifidase following dosing.
Imlifidase Pharmacokinetics (tmax) | From pre-dose imlifidase up to Day 15
  tmax = Time point for maximum observed plasma concentration of imlifidase following dosing
Imlifidase Pharmacokinetics (t1/2) | From pre-dose imlifidase up to Day 15
  t1/2 = Terminal half-life of imlifidase.
Imlifidase Pharmacokinetics (CL) | From pre-dose imlifidase up to Day 15
  CL = Clearance of imlifidase.
Imlifidase Pharmacokinetics (Vz) | From pre-dose imlifidase up to Day 15
  Vz = Volume of distribution during the elimination phase
Imlifidase Pharmacodynamic (PD) profile up to 9 days after imlifidase treatment | From pre-dose imlifidase up to Day 10
  PD is assessed as serum concentrations of intact IgG and its fractions following infusion.
Immunogenicity profile of imlifidase up to 5 years after imlifidase treatment | From pre-dose imlifidase up to 5 years
  Immunogenicity is assessed as serum concentration of anti-imlifidase IgG (ADA).
Proportion of patients with biopsy- and serology (DSA)-confirmed AMR up to 5 years after transplantation | From transplantation up to 5 years
  Banff scores (Loupy et al. 2020) will be used for biopsy evaluation.
Proportion of patients with biopsy confirmed cell-mediated rejection (CMR) up to 5 years after transplantation | From transplantation up to 5 years
  Banff scores (Loupy et al. 2020) will be used for biopsy evaluation.

OTHER OUTCOMES:
Safety assessed as proportion of patients with infusion related reactions within 48 hours of imlifidase infusion | From start of imlifidase infusion up to 48 hours
Safety assessed as proportion of patients with severe or serious infections within 30 days after imlifidase treatment | From start of imlifidase infusion up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Hansa Biopharma AB
Locations (4):
- HUS, Helsinki University Hospital, Helsinki, Finland
- Robert Debre University Hospital, Paris, France
- Hospital Unviersitari Vall d'Hebron, Nefrología Pediátrica, Barcelona, Spain
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loupy A, Haas M, Roufosse C, Naesens M, Adam B, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell LD, Clahsen-van Groningen MC, Demetris AJ, Dragun D, Duong van Huyen JP, Farris AB, Fogo AB, Gibson IW, Glotz D, Gueguen J, Kikic Z, Kozakowski N, Kraus E, Lefaucheur C, Liapis H, Mannon RB, Montgomery RA, Nankivell BJ, Nickeleit V, Nickerson P, Rabant M, Racusen L, Randhawa P, Robin B, Rosales IA, Sapir-Pichhadze R, Schinstock CA, Seron D, Singh HK, Smith RN, Stegall MD, Zeevi A, Solez K, Colvin RB, Mengel M. The Banff 2019 Kidney Meeting Report (I): Updates on and clarification of criteria for T cell- and antibody-mediated rejection. Am J Transplant. 2020 Sep;20(9):2318-2331. doi: 10.1111/ajt.15898. Epub 2020 May 28. PMID 32463180